CLINICAL TRIAL: NCT06354335
Title: Impact of a Major Organizational Change on Employee Productivity and Mental Health - a Register-based Cohort Study of the Relocation of a Large Danish Hospital in 2016-2019
Brief Title: Impact of a Major Organizational Change on Employee Productivity and Mental Health
Acronym: PRO-MENTA
Status: Active, not recruiting | Type: Observational
Sponsor: Aarhus University Hospital (Other)
Collaborators: University of Aarhus (Other); Herning Hospital (Other); Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Morten Vejs Willert, Senior researcher, Aarhus University Hospital
Other Study IDs: 1-16-02-62-20
Record Dates: First submitted 2024-03-26; First posted 2024-04-09 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Work Related Stress; Mental Health Issue; Work-related Illness
MeSH Terms: conditions — Occupational Stress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Employees: Persons employed at the hospital during 2011-2020
  Interventions: Other: Employees exposed to a major hospital reorganisation

INTERVENTIONS:
Other: Employees exposed to a major hospital reorganisation — Occupational exposure

SUMMARY:
The study investigates the short- and long-term impact of a major organizational change on employee health and productivity. Changes in organizations is a common aspect of modern work life in all sectors and public healthcare is no exception. However, emerging evidence suggests that organizational changes may be a potential stressor which can impact on employee well-being and contribute to stress-related health problems. Using a large-scale natural experiment, the overall aim of the study is to investigate the impact of a major organizational change that took place during 2016-19 on employee health and productivity. In addition, we aim to identify groups that may be at increased risk of experiencing negative consequences of the reorganization. These at-risk groups can in turn be candidates for extended preventive measures when planning future major organizational changes.

DETAILED DESCRIPTION:
The study relies solely on data from registries and the investigators have taken great care to ensure the validity of these data. Below the main principles and procedures applied are outlined. For the data delivered from the hospital Business Intelligence (BI) database the investigators performed interviews with representatives from each workplace. This was done to ensure that the information about when a workplace underwent the organizational change was accurate, but also what type of organizational change the workplace experienced, how the workplace was organized in terms of departments/wards, and the number of employees at the workplace.The validity of the data supplied by Statistics Denmark relies on the comprehensive procedures to ensure data integrity at Statistics Denmark. All datamanagement by the investigators has been performed in the Stata software package and all decisions are documented in program files (called "do-files" in Stata teminology) to ensure a complete revision trail from the delivered raw data to the dataset used for the final analyses. The investigators have performed extensive data checks, both by tabulations, codebooks, and visual inspection of the data. To ensure against data management errors done by a single investigator when writing the program/do-files, all coding performed in the datamanagement phase has been reviewed by at least one of the other researchers.

ELIGIBILITY:
Inclusion Criteria:

* All employees at the hospital during 2011-2020

Exclusion Criteria:

* Employees who, after being informed of the study, opted out of participation (N=70)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population covers all persons that have had an employment at the hospital during 2011-2020
Sampling Method: Non-Probability Sample
Enrollment: 31555 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Employee health measured by rate of absenteeism, use of health care services and redeemed drug prescriptions | 4 years in which the outcomes are measured monthly and form a time-series of observations for 2 years before and after workplace reorganization
  Employee health will be assessed monthly as rate absenteeism from work, use of general and mental health care services, and redeemed psychotropic drug prescriptions. The data are derived from a combination of company records and registries provided by Statistics Denmark

SECONDARY OUTCOMES:
Workplace productivity measured by number of patient contacts and medical procedures | 4 years in which the outcomes are measured monthly and form a time-series of observations for 2 years before and after workplace reorganization
  Workplace productivity is measured by the monthly number contacts and performed medical procedures. These are aggregated at the workplace level and derived from the Business Intelligence (BI) system of the hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Morten V Willert, PhD, Principal Investigator — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus, Central Jutland, Denmark

IPD SHARING:
Plan to Share IPD: No
The rules of Statistics Denmark prohibit the sharing of data from this study with other researchers.